CLINICAL TRIAL: NCT03315403
Title: Community-Acquired Pneumonia: lytA TArgeted Real Time Quantitative Polymerase chaIN Reaction for Improved Detection of Pneumococci (CAPTAIN)
Brief Title: Quantitative Polymerase Chain Reaction for Improved Detection of Pneumococci in CAP "CAPTAIN"
Acronym: CAPTAIN
Status: Completed | Type: Observational
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, W.G.Boersma, MD. PhD. Pulmonologist, Medical Center Alkmaar
Other Study IDs: 63200
Record Dates: First submitted 2017-10-03; First posted 2017-10-20 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Pneumonia, Pneumococcal; Community-acquired Pneumonia
Keywords: quantitative polymerase chain reaction; qPCR; autolysin; lytA; Pneumococcal pneumonia; Diagnostics; Community-acquired Pneumonia; Antibiotic resistance
MeSH Terms: conditions — Pneumonia, Pneumococcal; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of nasopharynx, oropharynx, saliva, sputum and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with CAP: Patients with a diagnosis of radiographically-confirmed CAP at the emergency department will undergo the usual diagnostics. For the study an extra nasopharynx sample, saliva sample and blood sample will be collected.
  A questionnaire will be filled in. LytA qPCR and cultures will be performed on samples of the upper respiratory tract (nasopahrynx, oropharynx, saliva, sputum if available)
  Interventions: Diagnostic Test: LytA targeted quantitative polymerase chain reaction (qPCR)
- Related controls: Of related controls a nasopharynx sample, oropharynx sample and saliva sample will be collected.
  A questionnaire will be filled in. LytA qPCR and cultures will be performed on samples of the upper respiratory tract (nasopahrynx, oropharynx, saliva)
  Interventions: Diagnostic Test: LytA targeted quantitative polymerase chain reaction (qPCR)
- Unrelated controls: Of unrelated controls a nasopharynx sample, oropharynx sample and saliva sample will be collected.
  A questionnaire will be filled in. LytA PCR and cultures will be performed on samples of the upper respiratory tract (nasopahrynx, oropharynx, saliva)
  Interventions: Diagnostic Test: LytA targeted quantitative polymerase chain reaction (qPCR)
- Patients with stable COPD: Of stable COPD patients a nasopharynx sample, oropharynx sample and saliva sample will be collected. And if available also a sputum sample.
  A questionnaire will be filled in. LytA qPCR and cultures will be performed on samples of the upper respiratory tract (nasopahrynx, oropharynx, saliva, sputum if available)
  Interventions: Diagnostic Test: LytA targeted quantitative polymerase chain reaction (qPCR)
- Patients with exacerbation of COPD: Of patients with a diagnosis of an exacerbation of COPD at the emergency department a nasopharynx sample, oropharynx sample and saliva sample will be collected apart from the usual diagnostics. If available also a sputum sample will be collected.
  A questionnaire will be filled in. LytA qPCR and cultures will be performed on samples of the upper respiratory tract (nasopahrynx, oropharynx, saliva, sputum if available)
  Interventions: Diagnostic Test: LytA targeted quantitative polymerase chain reaction (qPCR)

INTERVENTIONS:
Diagnostic Test: LytA targeted quantitative polymerase chain reaction (qPCR) — LytA qPCR and cultures will be performed on samples of the upper respiratory tract (nasopahrynx, oropharynx, saliva, sputum if available)

SUMMARY:
The purpose of this study is to evaluate the added diagnostic value of a quantitative polymerase chain reaction targeting the lytA gene in detecting pneumococci in patients with community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age 18 years or above;
* Presentation at the emergency department (ED);
* Working diagnosis of CAP at the ED with the presence of at least two of the following criteria:

  1. New or worsened coughing;
  2. Production of purulent sputum or change in sputum colour;
  3. Temperature >38.0 ⁰C or ≤36.0 ⁰C (tympanic);
  4. Auscultatory findings consistent with pneumonia, including rales, evidence of pulmonary consolidation (dullness on percussion, bronchial breath sounds, rales, or egophony), or both;
  5. White blood cell count of >10x10^9 cells/L or <4x10^9 cells/L or >15% bands;
  6. C-reactive protein level ≥30mg/L;
  7. Dyspnea, tachypnea, (>20 breaths per minute), or hypoxemia (arterial pO2 <60mmHg or peripheral O2 saturation <90%).
* New consolidation(s) on the chest radiograph or computed tomography (CT);
* No other explanation for the signs and symptoms;

Control group 1 - Related controls

* Being aged 18 years or above;
* Close relative of the patient: relative defined as living in the same house as the CAP patient or daily contact;
* Is at the hospital at the moment of inclusion of the CAP patient or is willing to come for testing within 7 days;

Control group 2 - Unrelated healthy individuals

* Being aged 18 years or above;
* Subject with a preoperative appointment with the anaesthiologist for a planned surgical procedure;
* Age matched to a included CAP patient (+-10 years);
* Time matched to a included CAP patient (up to 14 days after inclusion of the CAP patient);
* Gender matched to a included CAP patient.

Control group 3 - Patients with stable COPD

* Being aged 18 years or above;
* Diagnosis of COPD confirmed with spirometry (GOLD criteria 2017)(76);
* Stable disease.

Control group 4 - Patients with exacerbation of COPD

* Being aged 18 years or above;
* Diagnosis of COPD confirmed with spirometry (GOLD criteria 2017)(76);
* Diagnosis of exacerbation of COPD: defined as an acute event characterised by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medication (76).
* Presentation at emergency department with the suspicion of an exacerbation.

Exclusion Criteria:

In general:

* Recent pneumonia (< 1 month) or pneumonia in last 3 months with known pneumococcal aetiology with one of current diagnostics;
* Was included in the study group before;
* Not capable of understanding information needed to sign informed consent.

Patients:

* Aspiration pneumonia;
* Hospitalisation for two or more days in the last 14 days;
* History of cystic fibrosis.

For all control groups:

* Fits inclusion criteria for patient group;
* Present or recent hospitalisation (14 days);
* Fits inclusion criteria for patient group;
* Use of antibiotics in the last 14 days, including maintenance antibiotic therapy.

Control group 1 and 2 - Related healthy controls and unrelated healthy individuals

* Active infectious respiratory complaints defined as defined as two or more respiratory symptoms (cough, nasal congestion, runny nose, sore throat or sneezes);
* Temperature >38.0 ⁰C;
* Fits inclusion criteria for control group 3 or 4;
* Chronic pulmonary disease: COPD, asthma, cystic fibrosis, bronchiectasis.

Control group 3 - Patients with stable COPD

* Temperature >38.0 ⁰C;
* Stable disease;
* Fits inclusion criteria for control group 4;
* Recent exacerbation (<1 month) defined as increased respiratory symptoms with need of antibiotic and/or corticosteroid therapy;
* History of cystic fibrosis.

Control group 4 - Patients with exacerbation of COPD

* Current pneumonia;
* Recent exacerbation (<1 month) defined as increased respiratory symptoms with need of antibiotic and/or corticosteroid therapy;
* Fits inclusion criteria for control group 3;
* History of cystic fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient group: Adult patients ≥18 years with diagnosis of CAP at the emergency department (ED).
  Control groups (without CAP):
  * Related controls (inclusion at ED)
  * Unrelated healthy adults (inclusion at an outpatient preoperative appointment for any elective surgery)
  * Stable COPD patients (inclusion at outpatient clinic for pulmonary diseases)
  * COPD patients with an AECOPD (inclusion at ED)
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
qPCR diagnosed pneumococcal pneumonia | 1 day, day of inclusion
  Occurrence of qPCR proven pneumococcal pneumonia (CAP with S. pneumoniae detected by qPCR in at least one of the samples with a positive lytA qPCR and a DNA copy number above the determined cut-off value) using the cut-off value in at least one of the specimens at inclusion. The cut-off value will be determined in this study, see secondary objective.
Pneumococcal pneumonia with usual tests | 1 day, day of inclusion
  Occurrence of pneumococcal pneumonia proven by at least one of the routine microbiological tests (urine antigen test, blood culture and/or sputum culture). The difference between outcome measure 1 and 2 is the added diagnostic value.

SECONDARY OUTCOMES:
Number of DNA copies of S. pneumoniae in all lytA qPCR positive study subjects | 1 day, day of inclusion
  The number of DNA copies of every study subject with a positive qPCR will be determined. The optimal cut-off value will be determined to distinguish between colonisation and infection by comparing the number of DNA copies of controls with a positive lytA PCR and patients with a pneumococcal pneumonia proven by routine microbiological tests. This cut-off value will be used for outcome measure 1 to determine the amount of patients with an qPCR proven pneumococcal pneumonia.
Occurrence of positive lytA qPCR at 30 days after inclusion in CAP patients | 30 days
  Occurrence of positive lytA qPCR at 30 days after inclusion in CAP patients in the different samples: oropharynx, nasopharynx, saliva and sputum.
CURB-65 scores | 1 day, day of inclusion
  CURB-65 scores will be determined in CAP patients at moment of inclusion.
Procalcitonin | 1 day, day of inclusion
  Procalcitonin levels will be determined in CAP patients at moment of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Boersma, MD. PhD., Principal Investigator — Noordwest Ziekenhuisgroep
Locations (2):
- Netherlands (2):
  - Spaarne Gasthuis, Haarlem, North Holland
  - Noordwest Ziekenhuisgroep, Alkmaar